CLINICAL TRIAL: NCT03705689
Title: Validation BITSS Brussels Infant Stool Scale
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Yvan Vandenplas, head of Clinic, Universitair Ziekenhuis Brussel
Other Study IDs: 2018-365
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Validation of BITTS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: validation of Bitts — No intervention, observation of photographs of stool

SUMMARY:
validation of stool scale in toddlers

DETAILED DESCRIPTION:
objective : the Bristol stool form scale (BSFS) is inadequate for non-toilet trained children.

The Brussels Infant and Toddler Stool Scale (BITTS) was developed, consisting of 7 photograps of diapers containing stools of infants and toddlers. We aimed to evaluate inter-observer reliability of stool consistency assessment among parents, nurses and medical doctors using the BITTS.

Method :

In this multicenter cross-sectional study (2016-2017), Bitts photograps were rated according to the BSFS. The reliability of the BITTS was evaluated using the overall proportion of perfect agreement and the linearly weighted K statistic.

What is known :

* reliable assessment of stool consistency is important for evaluating children's defecation pattern and diagnosing gastrointestinal disorders.
* the reliability of the Bristol Stool Form Scale, developed for adults, has been debated for young children who are non-toilet trained and wear diapers

To get validation of the BITTS :

* a non-toilet trained child makes stool in diaper
* caregiver scores the aspect of the stool according to the BITTS
* caregiver takes a picture of the diaper
* after 1 monts she rescores the picture according to the BITTS

ELIGIBILITY:
Inclusion Criteria:pictures of diapers with stool of all childeren who are non-toilet trained

-

Exclusion Criteria:

* none

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: all children who are non-toilet trained
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the inter-observer reliability of stool consistency | 6months
  stool of a non-toilet trained child wuk be scired by a caregiver according to the BITTS. Then the caregiver takes a picter of this diaper with stool. After 1 month she rescores the picter according to BITTS

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No